CLINICAL TRIAL: NCT06660147
Title: PAOLA-1 Ancillary Study: Retrospective Validation of KELIM as a Predictive and Prognostic Factor for Maintenance Treatment With PARP Inhibitor After Platinum-Based Chemotherapy in First-Line Ovarian Cancer
Brief Title: Validation of KELIM as a Predictive/Prognostic Factor for Maintenance Treatment With iPARP in First-Line Ovarian Cancer
Acronym: KELI-PAOLA
Status: Recruiting | Type: Observational
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Other Study IDs: GINECO OV131
Record Dates: First submitted 2024-10-14; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer
Keywords: parp inhibitor; kelim; maintenance treatment
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This study aims to understand whether it is possible to predict the effectiveness of maintenance treatment with PARP inhibitors following first-line chemotherapy in ovarian cancer, and thus better target the patients who benefit from this treatment

ELIGIBILITY:
Inclusion Criteria: Patients randomised in the PAOLA-1 study -

Exclusion Criteria:Opposition to the use of your data for research purposes.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients randomised in the PAOLA-1 study :
  Patients with advanced FIGO stage IIIB-IV high grade serous or endometrioid ovarian, fallopian tube, or peritoneal cancer treated with standard first line treatment combining platinum based chemotherapy plus bevacizumab followed by a maintenance treatment by bevacizumab and Olaparib or placebo.
Sampling Method: Non-Probability Sample
Enrollment: 327 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
predictive and prognostic value of the KELIM score | 18 months
  To evaluate the predictive and prognostic value of the KELIM score in patients receiving maintenance treatment with a PARP inhibitor as part of the PAOLA-1 clinical trial.

CONTACTS AND LOCATIONS:
Locations (24):
- France (23):
  - ICO Paul Papin, Angers
  - Sainte-Catherine Institut du Cancer Avignon-Provence, Avignon
  - CHRU Besançon - Hôpital Jean Minjoz, Besançon
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU Grenoble-Alpes - Site Nord (La Tronche), Grenoble
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - Centre Azuréen de Cancérologie, Mougins
  - Hôpital Privé du Confluent, Nantes
  - Groupe Hospitalier Diaconesses - Croix Saint-Simon, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Curie, Paris
  - Clinique Francheville, Périgueux
  - HCL - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - Centre Eugène Marquis, Rennes
  - ICO - Centre René Gauducheau, Saint-Herblain
  - Oncopole Claudius Regaud - IUCT Oncopole, Toulouse
  - Clinique Pasteur, Toulouse
  - ICL - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Centre Hospitalier Princesse Grace, Monaco, Monaco